Date: June 29, 2023

# INFORMED CONSENT TO PARTICIPATE IN A RESEARCH PROJECT:

"Adherence to Different Exercise Interventions"

### INFORMED CONSENT TO PARTICIPATE IN A RESEARCH PROJECT:

"Adherence to Different Exercise Interventions"

#### INTRODUCTION

This form asks for your agreement to participate in a research project on adherence to exercise different interventions. Your participation involves attending 7 visits over 4-weeks to Cal Poly's Center for Health Research facilities. It is expected that your participation in the study visits will take approximately 4-5 hours over 4-weeks. The potential risks from this project are considered minimal. There are no direct benefits for participating in this study. You will be asked to participate in regular exercise over the 4-weeks. If you are interested in participating, please review the following information.

# PURPOSE OF THE STUDY AND PROPOSED BENEFITS

- The purpose of the study is to examine adherence to three different exercise interventions.
- There are no direct benefits associated with the study. These data are collected for research purposes only and are not clinical or diagnostic. These data may further our understanding of methods to increase adherence to exercise interventions.

# YOUR PARTICIPATION

- If you agree to participate, you will be asked to attend 7 visits over 4-weeks that will take approximately 4-5 hours. The visits are:
  - <u>Visit 1:</u> Informed Consent. You will be provided with a full description of the study and can ask any questions. At this time, you should inform the investigators of any other studies that you are participating in. If you are interested in participating in the study, you will be familiarized with the study visits. This visit will take approximately 1 hour.
  - <u>Visit 2:</u> Measure weight, height, and complete a demographic questionnaire, health history questionnaire, and physical activity questionnaire. You will be given a GENE-Active watch, which is an accelerometer and will be worn on your non-dominant wrist. You will be asked to keep the watch on for the entire study but may take it off at night when you sleep and when you shower. You will provide 3-days of baseline GENE-Active accelerometer data. This visit will take approximately 1 hour.
  - Visit 3: You will be randomized (you do not get to choose) to one of three exercise interventions: 1) walk intervention, 2) variety intervention, 3) progressive intervention. For the variety intervention, each week you will be asked to participate in a different exercise which will only include cycling, walking/jogging, yoga/Pilates, cross-training, and strength training. For the progressive intervention, the same exercises will be included but will be added to the list of options for you to participate in. You can choose from the list of exercise and can do as much or little of each exercise as you want (Here is an example: Week 1: yoga, Week 2: yoga and walking, Week 3: yoga, walking, and strength training, Week 4: yoga, walking, strength training, cross-training). The goal of each intervention is to exercise for at least 150 minutes per week. The exercise will not be supervised, and you will complete this on your own. This visit will take approximately 30 minutes.
  - O Visits 4-6: After each week you will meet with a study researcher that will download the watch accelerometer data, your weight will be measured, you will complete a physical activity diary, and you will be provided the next week exercise. These visits will take approximately 15 minutes each.

- O Visit 7. Final assessments of physical activity diary, watch accelerometer, and weight will be collected. We will also ask some open-ended questions on the acceptability of the intervention. This visit will take approximately 1 hour.
- There are no costs to participate in this study. There are no incentives for participating in this study.

#### PROTECTIONS AND POTENTIAL RISKS

- Please be aware that you are not required to participate in this research, refusal to participate will not involve any penalty or loss of benefits to which you are otherwise entitled, and you may discontinue your participation at any time without penalty or loss of benefits. Your participation is voluntary. If you are a student, your decision whether to participate will not have any effect on your academic status. Please feel free to ask questions at any time if there is anything you do not understand. Please be aware that you are not required to participate in this research, and you may omit any items you prefer not to answer on the questionnaires.
- The researcher may terminate your participation at any time. Possible reasons for removal are: if all or part of the study is stopped for any reason by the investigator or Cal Poly; if you are a student and participation in the study is adversely affecting your academic performance; if you fail to adhere to the requirements for participation established by the researcher.
- The possible risks or discomforts associated with participation in this study include potential physical, psychological, and social risk. During any type of exercise, especially strenuous exercise, there are slight health or physical risks, along with the possibility of fatigue and muscle soreness. These health risks are small in people with no prior history of cardiovascular, respiratory, or musculoskeletal disease or injury. Any ordinary fatigue or muscle soreness is temporary and usually lasts 24-96 hours. There are slight psychological and social risks of completing the questionnaires, and you may omit any question that you do not feel comfortable answering.
- Also, there is a slight risk of musculoskeletal injury with exercise, which is slighter higher in people that do not exercise regularly. However, the risk is much higher in people that perform high-impact sports like soccer, football, etc. As part of this study, you will not be asked to perform any contact sports that may increase the chance of a musculoskeletal injury.
- Your confidentiality will be protected as all information collected from you, including data sheets, watch accelerometer data, and questionnaire responses, will be coded, instead of using your name. We will use the codes, instead of your name, to analyze and report on the information learned from you, so that your information will be de-identified and cannot be traced. All paper records will be stored in a locked file that only project personnel will have access to. Online data will be encrypted, password protected and stored in the cloud using Cal Poly's Amazon Web Services.
- In any written or oral presentation of this research, your identity will be kept private. Records that identify you may be inspected by authorized individuals such as the Cal Poly Institutional Review Board, researchers on this study, or employees conducting peer review activities. Your agreement to participate indicates consent to such inspections and to the copying of excerpts of your records, if required by any of these representatives.
- All records will be kept in our database for 7 years after the date of the last participant completing
  the study, or the data may be destroyed if no longer in use before the 7 years. Your data may be
  shared with the broader scientific community or journals for publication upon request. Your data
  will be de-identified and they will not be allowed to have access to your name and other personal
  information.

- Identifying data will be removed from your private information and that, after such removal, the information could be used for future research studies or distributed to another researcher for future studies without additional informed consent.
- All study personnel have been trained at Cal Poly on the rights of human subjects, and they are familiar with the rules for handling personal information.

#### RESOURCES AND CONTACT INFORMATION

- If you should experience any negative outcomes from this research, please be aware that you may contact an appropriate referral source such as the Campus Health & Wellbeing if you are a student (805-756-1211), the researcher Dr. Todd Hagobian (805-756-7511) for assistance.
- This research is being conducted by Dr. Todd Hagobian, Professor in the Department of Kinesiology and Public Health at Cal Poly, San Luis Obispo, and Dr. Adam Seal, Postdoctoral Research Fellow in the Department of Kinesiology and Public Health at Cal Poly, San Luis Obispo. If you have questions regarding this study or would like to be informed of the results when the study is completed, please contact Dr. Hagobian at <a href="mailto:thagobia@calpoly.edu">thagobia@calpoly.edu</a> or 805-756-7511, or Dr. Adam Seal at <a href="mailto:adseal@calpoly.edu">adseal@calpoly.edu</a> or 805-756-2545.
- If you have concerns regarding the way the study is conducted, you may contact Dr. Michael Black, Chair of the Cal Poly Institutional Review Board, at (805) 756-2894, mblack@calpoly.edu, or Ms. Trish Brock, Director of Research Compliance, at (805) 756-1450, pbrock@calpoly.edu.

# AGREEMENT TO PARTICIPATE

If you are 18 or older and agree to voluntarily participate in this research project as described, please indicate your agreement by signing below. Please retain a copy of this form for your reference and thank you for your participation in this research.

| Yes, I agree to participate. | |
|------------------------------|------|
| Signature of Volunteer | Date |
| Signature of Researcher | Date |